CLINICAL TRIAL: NCT05558735
Title: Contribution of Canine Detection in the Diagnostic Strategy of High-risk Prostate Cancer
Brief Title: Contribution of Canine Detection in the Diagnostic Strategy of High-risk Prostate Cancer (Prostate-K9-Detect)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220569
Record Dates: First submitted 2022-09-15; First posted 2022-09-28 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-09

CONDITIONS: High-risk Prostate Cancer
Keywords: prostate cancer; canine detection; the dog's sense of smell
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: The case group is composed of Adult male with a positive biopsy (Gleason score greater than or equal to 7)
  Interventions: Other: urine collection; Other: canine detection
- control group: The control group is made up of adult men performing a biopsy whose Gleason score is less than or equal to 6.
  Interventions: Other: urine collection; Other: canine detection

INTERVENTIONS:
Other: urine collection — urine collection as part of the care and usual follow-up in the context of suspected prostate cancer
Other: canine detection — urine sample will be placed in a detection cone to be sniffed by 6 trained dogs

SUMMARY:
The sense of smell allows both humans and dogs to carry out a chemo-sensory analysis of their environment. Volatile organic compounds enter the nasal cavities and bind to receptors in the nasal mucosa. Neuroepithelium cells perform chemoelectric transduction of olfactory information. The latter is supported by one of the fibers of the olfactory nerve which crosses the cribriform plate of the ethmoid to arrive in the olfactory bulb of the brain. Incorporating this information can lead to behavioral responses. The dog has a sense of smell 100,000 times more sensitive than humans, it is able to detect one particle among 1 trillion. The use of detection dogs involves learning the behavioral response to an olfactory stimulus. Prostate cancer represents 25% of male cancers, it is the second deadliest cancer in France with 10,000 deaths per year. Diagnosis of prostate cancer requires a Prostate Specific Antigen (PSA) blood test and a digital rectal examination. In the event of an abnormality in one of these parameters, a prostate MRI is indicated, supplemented by prostate biopsies in the event of an abnormal MRI. However, one situation remains open to discussion: what should be done when faced with a normal MRI despite an abnormal PSA level or digital rectal examination? In this situation and according to current recommendations, the practitioner has the choice between performing prostate biopsies, i.e. an invasive procedure with a high risk of being negative, and simple monitoring, this time with the risk of missing the diagnosis of prostate cancer. Several studies have shown the effectiveness of dogs in detecting very specific volatile organic compounds. Can the investigators train them to detect the catabolites of prostate tumours?

DETAILED DESCRIPTION:
"The purpose of this study is to validate the diagnostic aid performance of canine detection of high-risk prostate cancers (Gleason score 7 or more) by comparing it to prostate MRI with respect to the results of biopsies of the prostate, then to integrate this test into the current diagnostic strategy for prostate cancer.

We will carry out a descriptive observational prospective case-control study at the Bichat-Claude Bernard and Henri Mondor hospitals (France) in routine care in adult patients suspected of prostate cancer and having an indication for the realization of a urine sample, an MRI prostate cancer and prostate biopsies.

The patient journey will be as follows :

During the initial visit (V1), patients suspected of prostate cancer (pathological digital rectal examination, PSA > 4) are informed about the study. They can entrust their non-objection to participate in the study now, or return during a new visit (V2) after a reflection period of 2 to 6 weeks.

Each patient completed a clinical information questionnaire. A 60 ml urine sample is taken, part of which is used to perform the ECBU necessary for performing prostate biopsies. The remainder of the sample is used for research.

The next visit (V3) is that of performing prostate biopsies, which provide the diagnosis of certainty on the presence or absence of prostate cancer. In the meantime, the patient performed an MRI of the prostate. All of these interventions are part of the usual management of patients suspected of prostate cancer. This visit is followed by the comparison of the results of canine detection and prostate MRI with the results of prostate biopsies.

The last visit (V4) is a one-year follow-up visit. A new PSA assay and a digital rectal examination will be performed as part of the usual care.

The patients included in our study require a urine sample as part of their therapeutic management.

Part of this urine will be collected for our study, it will be frozen and then transported to the veterinary school of Maisons-Alfort.

Our research is divided into 2 phases:

* The validation phase, consisting of evaluating the diagnostic aid performance of canine olfaction for the diagnosis of prostate cancer in comparison to prostate MRI.
* The last phase of clinical interest, aimed at integrating canine olfaction into the current diagnostic strategy for prostate cancer, in particular in the case of negative MRI.

The sensitivity of canine olfactory detection will be calculated by dividing the number of patients marked by dogs among the patients diagnosed with high-risk prostate cancer from the biopsy.

The sensitivity of detection by MRI will be calculated by dividing the number of patients for whom the MRI indicated the presence of high-risk prostate cancer among the patients diagnosed with high-risk prostate cancer from the biopsy.

The 95% confidence intervals will be calculated using Jeffrey's method. The two calculated sensitivities will be compared using McNemar's statistical test.

The specificity of canine olfactory detection will be calculated by dividing the number of patients not marked by dogs among the patients who did not have high-risk prostate cancers diagnosed from the biopsy.

The specificity of detection by MRI will be calculated by dividing the number of patients for whom the MRI did not indicate the presence of high-risk prostate cancer among the patients whose biopsy did not indicate the presence of high-risk prostate.

The 95% confidence intervals will be calculated using Jeffrey's method. The two calculated specificities will be compared using McNemar's statistical test.

The concordance assessment scale quantified by Kappa from Landis and Koch will be used to assess the degree of concordance between the two methods (MRI, canine detection) and the biopsy.

This study will:

* Assess the diagnostic capacity of canine detection of prostate cancer in the event of a negative MRI.
* To validate a diagnostic score for prostate cancer including canine detection.
* Identify effluvia in the urine characteristic of prostate cancer.
* Assess the link between the PSA blood level and the concentration of volatile organic compounds in the urine.
* Evaluate the influence of subjects' lifestyle on the diagnostic capacity of canine detection of prostate cancer.
* Evaluate the influence of the grade of severity of prostate cancer on the diagnostic capacity of prostate cancer of canine detection.

The study respects the measures put in place to deal with the COVID-19 epidemic."

ELIGIBILITY:
"Inclusion criteria :

* Older than 18 years old
* Requiring the realization of a collection of urine from the framework of their care
* Requiring a PSA blood test, prostate MRI and prostate biopsies in the framework of their care

Exclusion criteria :

* Absence of signed informed consent
* People who do not speak French
* Persons whose general condition does not allow to participate in the study
* Protected populations: under guardianship or under curatorship
* Persons deprived of their liberty by a judicial or administrative decision
* Persons receiving care psychiatric
* Absence of affiliation to a pension scheme social Security"

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male with a positive biopsy (Gleason score greater than or equal to 7)
Sampling Method: Probability Sample
Enrollment: 183 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
"The primary outcomes measures are the sensitivity (Se) and specificity (Sp) of canine detection for the diagnosis of prostate cancer and the Kappa concordance coefficient. " | 24 months
  The Se, the Sp and the kappa coefficient will be calculated for each diagnostic method (MRI and canine detection). The definitive diagnosis will be given by the results of the prostate biopsies.

SECONDARY OUTCOMES:
Calculate the Kappa coefficient quantifying the concordance between canine detection and biopsy, first among patients with negative MRI then among patients with positive MRI. | 24 months
Show that the percentage of marking of the dog when the MRI is negative and the biopsy positive is significantly greater than 50% (correct marking by simple chance). | 24 months
Compare the diagnostic score obtained using all the examinations carried out when prostate cancer is suspected (assay of the PSA level, digital rectal examination, MRI, prostate biopsy) with the score obtained by adding canine detection. | 24 months
  Each outcome measures will be transformed into a binary measurement in order to be able to create a diagnostic score. A PSA level greater than 4ng/mL is worth 1, while if it is less than 4ng/mL, the value 0 will be attributed to the patient. The presence of a nodule on the digital rectal examination is worth 1, while the absence of a nodule is worth 0. The presence of a target zone on the MRI is worth 1 while the absence of a target zone is worth 0. Marking by the dogs is worth 1 while non-marking is worth 0. The score therefore varies between 0 and 3 without the intervention of the dog and between 0 and 4 by integrating the dog. We will then compare the sensitivities and specificities obtained with these two scores to that of the biopsy, the objective being to determine whether the dog has an interest in the current diagnostic protocol.
Perform a mass spectrometry examination on samples from the "case" group | 24 months
  The objective is to determine which volatile organic compounds are present in the urine, allowing the dogs to differentiate the urine of a healthy patient from the urine of a patient suffering from prostate cancer. We will analyze the urine of some patients with prostate cancer using a mass spectrophotometer.
"Compare the canine detection performances of prostate cancer (Se and Sp) according to different parameters of the patient's lifestyle, according to the different grades of cancer, and according to breeds and ages of dogs." | 24 months
"Compare the performance of canine detection of prostate cancer (Se and Sp) with detection performance of prostate cancer by measuring the blood PSA level." | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Hermieu Jean-François, Surgeon, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat - Claude-Bernard, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided